CLINICAL TRIAL: NCT02655393
Title: A Single (Part A) and Multiple (Part B) Dose Study of AMAZ-02, a Food Derived Ingredient to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Profile in Healthy Elderly Subjects
Brief Title: A Single and Multiple Dose Study of AMAZ-02 to Evaluate Safety and Pharmacokinetics in Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 15.02.AMZ; OP095615.AMA - OP095715.AMA (Other: Amazentis SA)
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Aging; Mitochondrial Dysfunction; Muscle Function
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Mitopure 250 mg single dose (Experimental): single dose of Mitopure soft gel capsules at 250 mg dose, n=8 subjects (6 Active, 2 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 500 mg single dose (Experimental): single dose of Mitopure soft gel capsules at 500 mg dose, n=8 subjects (6 Active, 2 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 1000 mg single dose (Experimental): single dose of Mitopure soft gel capsules at 1000 mg dose, n=8 subjects (6 Active, 2 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 2000 mg single dose (Experimental): single dose of Mitopure soft gel capsules at 2000 mg dose, n=8 subjects (6 Active, 2 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 500 mg single dose-Food Effect (Experimental): single dose of Mitopure admixed in yoghurt at 500 mg dose, n=8 subjects (6 Active, 2 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 1000 mg single dose-Food Effect (Experimental): single dose of Mitopure admixed in yoghurt at 1000 mg dose, n=8 subjects (6 Active, 2 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 250 mg multiple dose (Experimental): Repeated 28 day dosing of Mitopure soft gel capsules at 250 mg dose, n=12 subjects (9 Active, 3 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 500 mg multiple 28 day dose (Experimental): Repeated 28 day dosing of Mitopure soft gel capsules at 500 mg dose, n=12 subjects (9 Active, 3 Placebo)
  Interventions: Dietary Supplement: Mitopure
- Mitopure 1000 mg multiple 28 day dose (Experimental): Repeated 28 day dosing of Mitopure soft gel capsules at 1000 mg dose, n=12 subjects (9 Active, 3 Placebo)
  Interventions: Dietary Supplement: Mitopure

INTERVENTIONS:
Dietary Supplement: Mitopure

SUMMARY:
Part A:

The study is a double-blind, randomized, single ascending doses, study in 24 healthy elderly male and female volunteers. Each subject will be randomized for two subsequent doses in three cohorts.

Part B:

The study is a double-blind, randomized, multiple ascending doses study in 36 healthy elderly male and female volunteers. Subjects will be randomized to receive study product or placebo for 28 days.

DETAILED DESCRIPTION:
Part A: Single Ascending Dose study of AMAZ-02 with 3 cohorts (each cohort n=8 subjects, total n=24 subjects). Cohorts undergo two periods of single dose intervention separated by 3 week washout. Adverse events, clinical biochemistry for safety assessment and plasma and urine collected for pharmacokinetic measurement for parent and metabolite levels in circulation.

Part B: Multiple Ascending Dose study with 3 cohorts (each cohort n=12 subjects, total n=36 subjects). 28 day administration with AMAZ-02 for safety, PK and PD assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female elderly subject, aged between 61 and 85 years inclusive;
2. Non-smoker subject or smoker of not more than 5 cigarettes a day;
3. Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive;
4. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination);
5. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

   * 95 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 160 mmHg,
   * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 95 mmHg,
   * 50 bpm < HR < 80 bpm,
   * Or considered NCs by investigators;
6. Normal ECG recording on a 12-lead ECG at the screening visit:

   * 120 < PR < 220 ms,
   * QRS < 120 ms,
   * QTcf < 430 ms for male and < 450 ms for female,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCS by investigators;
7. Laboratory parameters within the normal range of the laboratory (haematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator;
8. Normal dietary habits;
9. Demonstrate sedentary behaviour defined as having an activity category of 1 as assessed by the International Physical Activity Questionnaire (IPAQ). Activity level is < 600 MET (metabolic equivalent unit - minutes per week and limited to light intensity activities.
10. Accept to refrain consuming certain foods and supplements at least two weeks before inclusion.
11. Comprehension of the nature and purpose of the study and ability to communicate in person and by telephone in a manner that allows all protocol procedures to be carried out safety and reliably in the opinion of the investigative site staff
12. Ability to take up to 8 capsules of study medication
13. Signing a written informed consent prior to selection;
14. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease;
2. Frequent headaches and / or migraine, recurrent nausea and / or vomiting;
3. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position;
4. Blood donation (including in the frame of a clinical trial) within 2 months before administration;
5. General anaesthesia within 3 months before administration;
6. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician;
7. Lactose intolerance, milk protein or soy allergy.
8. Inability to abstain from intensive muscular effort;
9. No possibility of contact in case of emergency;
10. Use of any of the prohibited medications as detailed in the concomitant medication section
11. History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day);
12. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day);
13. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests;
14. Positive results of screening for drugs of abuse;
15. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
16. Exclusion period of a previous study;
17. Administrative or legal supervision;
18. Subjects should not have participated in previous clinical trials in the last 3 months and received compensation beyond a certain approved and predefined limit

Ages: 61 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 6 weeks

SECONDARY OUTCOMES:
Plasma concentrations of AMAZ-02 and its metabolites over time and maximal plasma concentration (Cmax) | 6 weeks
Exposure to AMAZ-02 measured as area under the curve (AUC) | 6 weeks
Half-live (t 1/2) of AMAZ-02 and its metabolites | 6 weeks
Cmax of AMAZ-02 and its metabolites in urine | 6 weeks
AUC of AMAZ-02 and its metabolites in urine | 6 weeks
Gene expression for mitochondrial biomarkers in PBMC | 6 weeks
Gene expression for mitochondrial biomarkers in muscle tissue | 6 weeks
Blood Lipid Profile | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Latreille-Barbier, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France

REFERENCES:
- [Background] Andreux PA, Blanco-Bose W, Ryu D, Burdet F, Ibberson M, Aebischer P, Auwerx J, Singh A, Rinsch C. The mitophagy activator urolithin A is safe and induces a molecular signature of improved mitochondrial and cellular health in humans. Nat Metab. 2019 Jun;1(6):595-603. doi: 10.1038/s42255-019-0073-4. Epub 2019 Jun 14. PMID 32694802